CLINICAL TRIAL: NCT03275038
Title: Comparing Effects and Neural Mechanisms of Tai Chi and Light-to-Moderate Intensity on the Prevention of Leukoaraiosis and Declines in Brain, Physical, and Psychological Functions in Middle-aged and Older Adults With Cardiovascular Risks
Brief Title: Comparing Effects and Neural Mechanisms of Tai Chi and Light-to-Moderate Intensity Aerobic Exercises
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201612213RINB
Record Dates: First submitted 2017-08-30; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-03

CONDITIONS: Physical Activity
Keywords: Neuroimage; Training; Aging; Brain; Cardiovascular risks
MeSH Terms: conditions — Motor Activity | interventions — Aquatic Therapy; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Maintain the original life style
- Tai-Chi exercise group (Experimental): Receive three one-hour Tai Chi exercise sessions weekly for 24 weeks, supervised for the first 12 weeks and unsupervised for the next 12 weeks
  Interventions: Behavioral: Tai-Chi exercise
- Aerobic exercise group (Experimental): Receive three one-hour aerobic exercise sessions weekly for 24 weeks, supervised for the first 12 weeks and unsupervised for the next 12 weeks
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Tai-Chi exercise — Behavioral: Tai-Chi exercise
  Arms: Tai-Chi exercise group
Behavioral: Aerobic exercise — Behavioral: Aerobic exercise
  Arms: Aerobic exercise group

SUMMARY:
In this three-year project, investigators will target on sedentary middle-aged and older adults with cardiovascular risks, prescribe 24-week Tai Chi or aerobic exercises and examine:

1. Whether both exercises are effective to reduce cardiovascular risks, prevent leukoaraiosis and associated declines in physical and psychological functions at Week 12 and 24;
2. Will Tai Chi exercises be more effective on improving psychological health (cognition, psychological well-being, and exercise self-efficacy) than aerobic exercises at Week 12 and 24? If yes, are these effects mediated by specific brain structural and functional mechanisms?
3. Will aerobic exercises be more effective on improving physical health (motor functions, physical fitness, and heart rate variability) than Tai Chi exercises at Week 12 and 24? If yes, are these effects mediated by other specific brain structural and functional mechanisms?
4. After 12 and 24 weeks of Tai Chi and aerobic exercises, what are the relationships between reduction of cardiovascular risks and changes in brain structure and functions?

An assessor-blind randomized controlled clinical trial will be used. Based on known effect size of Tai Chi exercises on cognitive function (please refer to CM03, pages 9-10), 120 sedentary middle-aged and older adults with cardiovascular risks will be recruited and randomly assigned to the Tai Chi, Aerobic, or Control (usual care) group. The Tai Chi and Aerobic groups will receive three one-hour exercise sessions weekly for 24 weeks, supervised for the first 12 weeks and unsupervised for the next 12 weeks. The Control group will maintain the original life style. Clinical measures of cardiovascular risks and blood markers, brain structures and functional images, psychological (cognitive, psychological well-being and exercise self-efficacy) and physical (motor functions, physical fitness, and heart rate variability) functions will be collected at baseline, Week 12, and Week 24 to compare differences among the three groups across the three time points. Investigators will also examine the interrelationships of changes in brain structural and functional organization with changes in other measures, in an effort to understand the neural mechanisms of exercise effects.

DETAILED DESCRIPTION:
Leukoaraiosis prevails in middle-aged and older adults with cardiovascular risks. People with more severe leukoaraiosis would have greater risks for stroke, dementia, and disability. Tai Chi and aerobic exercises both can reduce cardiovascular risks; however, it remains unknown whether these two types of exercises also could prevent leukoaraiosis and associated declines in physical and psychological functions. In particular, would Tai Chi, a form of mind-body exercise, be more effective than aerobic exercises on improving psychological health with specific underlying brain structural and functional mechanisms? Would aerobic exercise be more effective than Tai Chi on improving physical healthy with different underlying brain structural and functional mechanisms?

Therefore, in this three-year project, investigators will target on sedentary middle-aged and older adults with cardiovascular risks, prescribe 24-week Tai Chi or aerobic exercises and examine:

1. Whether both exercises are effective to reduce cardiovascular risks, prevent leukoaraiosis and associated declines in physical and psychological functions at Week 12 and 24;
2. Will Tai Chi exercises be more effective on improving psychological health (cognition, psychological well-being, and exercise self-efficacy) than aerobic exercises at Week 12 and 24? If yes, are these effects mediated by specific brain structural and functional mechanisms?
3. Will aerobic exercises be more effective on improving physical health (motor functions, physical fitness, and heart rate variability) than Tai Chi exercises at Week 12 and 24? If yes, are these effects mediated by other specific brain structural and functional mechanisms?
4. After 12 and 24 weeks of Tai Chi and aerobic exercises, what are the relationships between reduction of cardiovascular risks and changes in brain structure and functions?

An assessor-blind randomized controlled clinical trial will be used. Based on known effect size of Tai Chi exercises on cognitive function (please refer to CM03, pages 9-10), 120 sedentary middle-aged and older adults with cardiovascular risks will be recruited and randomly assigned to the Tai Chi, Aerobic, or Control (usual care) group. The Tai Chi and Aerobic groups will receive three one-hour exercise sessions weekly for 24 weeks, supervised for the first 12 weeks and unsupervised for the next 12 weeks. The Control group will maintain the original life style. Clinical measures of cardiovascular risks and blood markers, brain structures and functional images, psychological (cognitive, psychological well-being and exercise self-efficacy) and physical (motor functions, physical fitness, and heart rate variability) functions will be collected at baseline, Week 12, and Week 24 to compare differences among the three groups across the three time points. Investigators will also investigate the interrelationships of changes in brain structural and functional organization with changes in other measures, in an effort to understand the neural mechanisms of exercise effects.

Results of this study will not only provide scientific evidence basis for clinical decision-making of using exercise approaches to prevent the development of leukoaraiosis and its negative health impact in middle-aged and older adults with cardiovascular risks, but also reveal the underlying neural mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 45 and 80 years old
2. Literacy
3. With cardiovascular risks, defined as having hypertension (defined as resting systolic BP≧140 mmHg or resting diastolic BP≧90 mmHg, or receiving antihypertensive medication), diabetes mellitus (defined as taking oral antidiabetics or insulin or fasting plasma glucose being ≥100 mg/dL), dyslipidemia (defined as receiving lipid-lowering medication and diet therapy or total cholesterol > 200 mg/dL or triglyceride > 150 mg/dL (Lan et al., 2008)), or a combination of two or three of these risks
4. Being physically inactive (defined as being engaged in physical activities for less than a total of 90 minutes per week) in recent one year
5. Have no prior experiences with Tai Chi, yoga, chi gung, or other meditative forms of exercises
6. No expectation of the need of changing medication in the following 8 months from the physicians

Exclusion Criteria:

1. Having any contraindications for fMRI (e.g., claustrophobia and indwelling metals or implanted devices)
2. Serious or uncontrolled cardiac or metabolic conditions (e.g., unstable angina, serious cardiac arrhythmias, heart failure, hypertrophic cardiomyopathy, severe aortic or carotid stenosis, pulmonary embolus or infarction, resting systolic BP ≥ 180 mmHg, resting diastolic BP ≥ 110 mmHg, fasting plasma glucose ≥ 300 mg/dL)
3. Severe renal failure
4. Symptoms or history of neurological diseases, including transient ischemic attack
5. Severe musculoskeletal disorders which would affect their mobility
6. Dementia or inability to follow instructions
7. Psychiatric disorder
8. Having contraindications for doing exercises (e.g., resting systolic BP ≥ 180 mmHg, resting diastolic BP ≥ 110 mmHg, fasting plasma glucose ≥ 300 mg/dL, hypoglycemia (plasma glucose ≤ 70 mg/dL) after exercises, and postural hypotension (BP drop ≥ 20 mmHg when changing postures)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-08-31 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Brain functional activation and structure imaging | up to 6 months
  fMRI activation patterns and white and gray matter changes of the brain

SECONDARY OUTCOMES:
Physical Activity Scale for the Elderly | up to 6 months
  assess daily physical activity
Geriatric Depression Scale short-form | up to 6 months
  assess emotional status
Mindfulness Attention Awareness Scale | up to 6 months
  assess mindfulness and attention
The AD8 scale | baseline
  A brief informant interview to detect dementia

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fang Tang, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Collage of Public Health, Taipei, Zhongzheng, Taiwan